CLINICAL TRIAL: NCT02306226
Title: Symetis ACURATE Neo™ Valve Implantation Using TransFemoral Access: SAVI TF Registry
Brief Title: Symetis ACURATE Neo™ Valve Implantation SAVI TF Registry
Acronym: SAVI TF
Status: Completed | Type: Observational
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Other Study IDs: 2013-05
Record Dates: First submitted 2014-09-02; First posted 2014-12-03 (Estimated); Last update posted 2018-03-19 (Actual); Status verified 2018-03

CONDITIONS: Aortic Stenosis
Keywords: TAVI; Aortic stenosis; Transcatheter aortic valve replacement; Transcatheter aortic valve implantation; Transfemoral access
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

SUMMARY:
Post-market registry aimed at further evaluating the safety and performance of the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System in patients with severe aortic stenosis treated with the commercialized device

DETAILED DESCRIPTION:
The SAVI TF is s single arm, multicenter, non-randomized and open registry. The purpose of this registry is to collect and monitor ongoing safety and performance data from commercial use of the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System.

The ACURATE neo™ and its Transfemoral Delivery System are intended for use in minimally invasive, transcatheter aortic valve replacement (TAVR) using transfemoral access in patients presenting with severe aortic valve stenosis.

The primary objective is to further evaluate the safety and performance of the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System in the first 1000 consecutive patients with severe aortic stenosis treated with the newly marketed device.

The secondary objective is to evaluate adverse events and device performance of the newly marketed device.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is included in the registry if eligible for transcatheter treatment of severe aortic stenosis with the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System as per the Instructions for Use
2. Patient is willing to participate in the study, provides signed Informed Consent/Data Authorization Form and authorizes the sharing of data in the registry
3. The subject and treating physician agree the subject will return for all required post-procedure follow-up visits

Exclusion Criteria:

1. Patients are excluded from the registry if they are not eligible for transcatheter treatment of severe aortic stenosis with the ACURATE neo™ Aortic Bioprosthesis and ACURATE TF™ Transfemoral Delivery System as per the Instructions For Use.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: As the ACURATE neo™ is approved for use to treat patients with severe aortic stenosis, the inclusion criteria are broad in order to allow the device to be used in an all-comers population and following the Instructions For Use.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-09; Primary Completion 2016-05 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Rate of all-cause mortality | 30 days

OTHER OUTCOMES:
Rate of clinical endpoints (VARC 2) | Procedure, 7 days or discharge (whichever occurs first), 30 days, 12 months
  * Mortality
  * Stroke
  * Myocardial infarction
  * Bleeding complication
  * Acute kidney injury
  * Vascular complication
  * Conduction disturbances and arrhythmia
  * Other TAVI-related complications
Procedural success | Post-implantation
  Procedural success defined as ACURATE neo™ implanted in intended location with:
  * Valve insufficiency < Grade 3
  * Mean aortic gradient < 20 mmHg
  * EOA ≥ 1.0 cm2
  * No valve-in-valve or conversion to surgery performed
  * No intra-procedure mortality
Device success | 7 days or discharge (whichever occurs first), 12 months
  Device success as defined as:
  * ACURATE neo™ implanted in intended location
  * No impingement of the mitral valve
  * Normal coronary blood flow
  * Valve insufficiency < Grade 3
  * Mean gradient < 20mmHg
  * EOA ≥ 1.0 cm2
  * No valve-in-valve or conversion to surgery performed
Functional improvement from baseline as per NYHA Functional Classification at 7 days or discharge (whichever occurs first), 30 days and 12 months follow-up | 7 days or discharge (whichever occurs first), 30 days and 12 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Helge Möllmann, Prof., Principal Investigator — Kerckhoff Klinik